CLINICAL TRIAL: NCT06435403
Title: SARS-CoV-2 Specific Antibody Responses and Impact for COVID-19 Disease in Health Care Worker and Community Members From Ethiopian Related to Natural SARS CoV-2 Infection and COVID-19 Vaccination
Brief Title: SARS-CoV-2 Specific Antibody Responses and Impact for COVID-19 Disease in Ethiopia
Acronym: CoVICIS
Status: Recruiting | Type: Observational
Sponsor: Michael Hoelscher (Other)
Collaborators: St. Paul's Hospital Millennium Medical College, Ethiopia (Other); Jimma University (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Director, Division of Infectious Diseases and Tropical Medicine, LMU Munich, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: ETH-02
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: SARS CoV 2 Infection; COVID-19 Breakthrough; COVID-19 Recurrent
Keywords: COVID-19; Seroepidemiologic Studies; Longitudinal Studies; Ethiopia / epidemiology; SARS-CoV-2
MeSH Terms: conditions — COVID-19; COVID-19 breakthrough infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 (N=300): SARS-CoV-2 anti-nucleocapsid positive, vaccinated
- Group 2 (N=300): SARS-CoV-2 anti-nucleocapsid positive, not vaccinated
- Group 3 (N=300): SARS-CoV-2 anti-nucleocapsid negative, vaccinated
- Group 4 (N=100): SARS-CoV-2 anti-nucleocapsid negative, not vaccinated

SUMMARY:
In this study we aim to characterize SARS CoV-2 strain specific immune response (SARS-CoV-2 Spike IgG) in health care workers and general populations at the Jimma Medical Center and the St. Paul Hospital in Addis Ababa in association to clinical immune protection and Covid-19 disease. Participants, stratified by SARS-CoV-2 infection and vaccination status, will be followed at 3-month intervals for a maximum of 2 years. Prevalence, incidence, and dynamics of SARS-CoV-2 specific antibodies as well as clinical assessments especially related to COVID-19 breakthrough disease in previously exposed/vaccinated participants will be performed. From a subset of selected participant blood sample, more in depth immunological analysis will be performed that include virus culture-based neutralization assays, antibody avidity assays, SARS-CoV-2 specific antibody epitope recognition using peptide arrays, and T-cell immunity assays (IGRA).

We also plan to analyze and model cost-effectiveness considerations related to adapted COVID-19 vaccine strategies, specifically if SARS-CoV-2 the costs for routine sero-diagnosis in high SARS-CoV-2 prevalent population prior to vaccination will impact the decision to vaccinate (no vaccination for low-risk populations or reduced vaccine dosing) and is cost-efficient. The study is largely exploratory, providing deeper insights in SARS-CoV-2 specific immune responses and interaction with SARS-CoV-2 viral variants.

DETAILED DESCRIPTION:
The COVID-19 pandemic has severely impacted health systems, interventions for infection control and resulting preventive public life restrictions. In a recent study, we determined high rates of previous SARS-CoV-2 infection in health care worker (over 70%) and communities in Ethiopia (up to 60%), with resulting potential natural acquired SARS-CoV-2 specific immunity. In contrast to the situation in Europe, the scale out of COVID-19 vaccination is however very low, and currently there is a scarcity of COVID-19 vaccines available all over Africa. Naturally acquired or vaccine induced SARS-CoV-2 immune responses have shown to protect against (severe) COVID-19 disease. However, immune responses are waning over time and new SARS-CoV-2 viral variants increasingly demonstrate immune escape properties. Correlates of clinical immune protections are currently investigated including binding SARS-CoV-2 spike IgG or neutralizing antibody levels, as well as cellular immune responses. However, threshold of immune protection are not yet defined that would guide the need of booster vaccinations, including for individuals with natural acquired immunity. There is evidence, that vaccination regimens in those individuals could be abbreviated to single shot booster, that would greatly economize challenged COVID-19 strategies in Africa.

The CoVICIS is a network of European and African researcher who collaborate on the overall objective to investigate SARS-CoV-2 specific immune response and correlates of immune protection in the context of circulating SARS-CoV-2 viral variants. In this affiliated study, we aim to investigate these outcomes in Ethiopian health care worker and community members throughout a longitudinal, prospective cohort study. Participants, stratified according to their SARS-CoV-2 infection and vaccination status, will be followed-up in 3-monthly intervals To characterize SARS CoV-2 strain specific immune response (SARS-CoV-2 Spike IgG) in health care workers and general populations stratified by previous (1) SARS CoV-2 exposure (SARS-CoV-2 anti-nucleocapsid antibody positive versus negative) and (2) vaccination status at the Jimma Medical Center (JMC) and the St. Paul Hospital in Addis Ababa in association to clinical immune protection and Covid-19 disease. Prevalence, incidence, and dynamics of SARS-CoV-2 specific antibodies as well as clinical assessments will be performed in 3-monthly intervals over a maximum period of 24 months.

At each study visits, immune responses including SARS-CoV-2 spike IgG and neutralizing antibody will be measured. In addition, SARS CoV-2-specific T cell responses will be studied in each of the study groups. COVID-19 disease or SARS-CoV-2 infections will be assessed throughout the study by clinical history, SARS-CoV-2 PCR diagnostics, and seroconversion of SARS-CoV-2 anti-nucleocapsid antibody testing as appropriate. In addition, more in-depth analysis will be performed in a subset of stored blood samples at collaborating specialized laboratories in Germany and Switzerland, including peptide array mapping, T-cell assays and affinity/avidity analysis against the ACE-II receptor. We further aim to characterize circulating SARS CoV-2 strains from PCR isolates in the context of investigated immune responses. Outcome results will be provided for computational analysis, integrating models for immune protection. Finally, we will explore the feasibility and cost-effectiveness of abbreviated single shot COVID-19 vaccination for individuals with pre-existing natural immunity to assess COVID-19 vaccine strategies that are especially applicable in African settings.

Findings from this study aim to help in guiding the current Covid-19 control strategy in Ethiopia. It might also give the first insight about the dynamics and level of antibodies produced against SARS-CoV-2 in the Ethiopian population.

ELIGIBILITY:
Inclusion criteria:

1. Adults, 18 years of above
2. Provision of oral as well as written informed consent
3. Available estimation of the period or the time-point when SARS-CoV-2 infection occurred (e.g. confirmed or highly suspected COVID-19 disease, SARS-CoV-2 anti-nucleocapsid seroconversion) (only applicable for participants included in group 1 and 2).
4. Employed/working in hospital (medical doctors, nurses/midwives, students, auxiliary personnel such as cleaner, runner, social worker) for HCW
5. Willingness to provide blood samples by venipuncture for serology and immunological characterization
6. Willingness to provide health information, report medical events and to performed SARS-CoV-2 diagnostics (swabs for PCR) in the case of suspected COVID-19 disease

Exclusion criteria:

1. Prisoners
2. Mentally disturbed persons
3. Persons for whom study participation will induce an unacceptable risk or burden as judged by the investigator (e.g. seriously sick persons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers (clinical staff, practicing medical interns, cleaners, guards, food handlers, and receptionists) at the two hospitals and potentially participants from the general urban population in Jimma and Addis Ababa will be included. N=500 participants at each site (N=1000 in total) will be stratified according to their SARS CoV-2 sero-s and Covid-19 vaccination status at inclusion into 4 groups. We aim to target at least 30% representation of HCW's, respectively community participants for each study group.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Difference of antibody levels between study groups by month 12 | 12 months
  Antibody levels will be compared between study groups by month 12
Proportion of participants with suspected clinically reported severe COVID-19 disease or evidence of SARS-CoV-2 exposure between study groups by month 12 | 12 months
  The proportion of participants with suspected clinically reported severe COVID-19 disease or evidence of SARS-CoV-2 exposure between study groups by month 12 will be compared
Proportion of SARS-CoV-2 breakthrough infections in previously exposed/vaccinated participants | 24 months
  The proportion of SARS-CoV-2 breakthrough infections in previously exposed/vaccinated will be compared

SECONDARY OUTCOMES:
Difference of antibody levels between groups by month 6, 18 and 24 | 24 months
  Antibody levels will be compared between study groups by month 6, 18, 24
Antibody levels after single 1st vaccination in previously infected persons | 24 months
  Antibody levels will be compared after single 1st vaccination in previously infected persons
Proportion of participants with suspected clinically reported severe COVID-19 disease or evidence of SARS-CoV-2 exposure between study groups by month 6, 18 and 24 | 24 months
  The proportion of participants with suspected clinically reported severe COVID-19 disease or evidence of SARS-CoV-2 exposure between study groups by month 6, 18 and 24 will be compared
Prevalence and distribution of circulating SARS-CoV-2 variants around baseline and during the study period | 24 months
  Prevalence and distribution of circulating SARS-CoV-2 variants around baseline and during the study period
Comparing costs related to SARS-CoV-2 anti-nucleocapsid diagnostics in relation to spared costs by abbreviated/not performed COVID-19 vaccine regimen | 24 months
  Comparing costs related to SARS-CoV-2 anti-nucleocapsid diagnostics in relation to spared costs by abbreviated/not performed COVID-19 vaccine regimen

OTHER OUTCOMES:
Difference of neutralizing antibodies in a subset of participants by study groups at baseline and subsequent time points | 24 months
  Comparing neutralizing antibodies in a subset of participants by study groups at baseline and subsequent time points
Recognition of SARS-CoV-2 specific peptide in a subset of participants by study groups at baseline and subsequent time points | 24 months
  Recognition of SARS-CoV-2 specific peptide in a subset of participants by study groups at baseline and subsequent time points
Determination of upper respiratory viral load in subjects with (re)infection | 24 months
  Determination of upper respiratory viral load in subjects with (re)infection

CONTACTS AND LOCATIONS:
Locations (2):
- Ethiopia (2):
  - Department of Microbiology Immunology and Parasitology, Addis Ababa
  - Jimma University, Jimma